CLINICAL TRIAL: NCT03946787
Title: EMDR Therapy in Relapse Prevention in Mood Episodes in Adolescents With Bipolar Disorder and History of Trauma: A Randomized Clinical Trial
Brief Title: EMDR in Adolescents With Bipolar Disorder and History of Trauma
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2018-0345
Record Dates: First submitted 2019-04-17; First posted 2019-05-13 (Actual); Last update posted 2019-05-13 (Actual); Status verified 2019-04

CONDITIONS: Bipolar Disorder
MeSH Terms: conditions — Bipolar Disorder | interventions — Eye Movement Desensitization Reprocessing; Therapeutics

STUDY DESIGN:
Intervention Model Description: 1. Group A: Treatment as Usual (TAU);
  2. Group B: TAU plus Eye Movement Desensitization and Reprocessing (EMDR) Therapy
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EMDR Therapy + TAU (Active Comparator): Patients will be submitted to 20 individual sessions of Eye Movement Desensitization and Reprocessing (EMDR) Therapy of 60 minutes each, combined to the Treatment as usual (TAU).
  It's an eight-step process aimed at the traumatic events, also used to address current situations that evoke emotional disturbances so they do not trigger more symptomatic reactions. In addition, it is helpful to assist the patient in developing the specific skills and behaviors required for a healthy functional life.
  Our group will adapt the EMDR protocol model specific for bipolar patients with a history of trauma, developed by Ahmann et al (2017), who applies EMDR in adults with Bipolar Disorder (BD) and history of trauma.
  Interventions: Other: Eye Movement Desensitization and Reprocessing (EMDR) Therapy; Other: Treatment as Usual
- TAU (Treatment as Usual) (Placebo Comparator): Patients will receive the Treatment as Usual. TAU will consist of the psychopharmacological approach appropriate to each patient according to the evaluation of a psychiatrist of childhood and adolescence's outpatient service. Patients are expected to be euthymic (or with subsyndromal symptoms) with the same medication for at least 3 months.
  Although the medications used by patients are relevant and taken into account in future analyzes, our group will not interfere with drug treatment. Thus, patients who require any type of drug intervention will be considered losses.
  Interventions: Other: Treatment as Usual

INTERVENTIONS:
Other: Eye Movement Desensitization and Reprocessing (EMDR) Therapy — The reprocessing and desensitization of each traumatic memory occurs in eight phases. In the first two phases, the therapist identifies targets and develops a treatment plan, enhances and develops personal resources, before working on traumatic memories. In stages 3 to 6, reprocessing and desensitization of memory is done. The patient focuses on the image of the event, negative beliefs and associated bodily sensations, while moving the eyes from side to side, following the therapist's fingers or other dual attention stimuli (eg, manual touch, auditory stimulation). Phases 7 and 8 are closing and reassessing, where the therapist determines if the memory has been processed properly.
  Other Names: EMDR Therapy
  Arms: EMDR Therapy + TAU
Other: Treatment as Usual — TAU will consist of the psychopharmacological approach appropriate to each patient according to the evaluation of a psychiatrist of childhood and adolescence's outpatient service.
  Other Names: TAU

SUMMARY:
In this research, EMDR protocol model specific for bipolar patients with a history of trauma, developed by Benedikt Ahmann et al (2017), who applies EMDR in adults with Bipolar Disorder (BD) and history of trauma will be adapted for adolescents. This protocol consists of a detailed survey of traumatic events, intervention and processing of these events according to the standard protocol developed by Shapiro.

The main hypothesis is that the use of EMDR in adolescents with BD and history of trauma, as a complement to the pharmacological treatment (Usual Treatment), would have beneficial effects in the course of the disease. Thus, the overall objective of this study is to examine whether EMDR therapy in adolescents with BD and history of traumatic events can reduce affective relapses within a 12-month period. In addition, improvement in biological markers related to BD is expected to be found when compared to the Usual Treatment. It is also expected that patients treated with EMDR will present a better neurocognitive functioning profile, assessed by means of a neuropsychological evaluation battery before and after the intervention, since recent studies show that the profile of humoral dysregulation, impulsiveness, difficulty in dealing with frustrations and social feedback in children and adolescents with BD is associated with poor cognitive control and executive function deficits.

DETAILED DESCRIPTION:
This will be a randomized controlled trial. Participants will be assigned to Eye Movement Desensitization and Reprocessing (EMDR) Therapy or Treatment as Usual (TAU) through block randomization. This process will be done using the program available at www. randomization.com.

In this study, EMDR Therapy will be applied in adolescents with BD and compared to the Usual Treatment. The neuropsychological profile of the patients will be evaluated before and after the interventions. In addition, the collection of the biological markers related to BD will be done by measuring the levels of salivary cortisol and serum levels of C-reactive protein (CRP), Brain Derived Neurotrophic Factor (BDNF), Interleukin (IL) - 1β, IL - 2, IL - 4, IL - 6, IL - 10, Interferon gamma (IFN-γ) and Tumor Necrosis Factor alpha(TNF-α) in these patients, since a study proposing the use of serological biomarkers for BD diagnosis concluded that the use of a single biomarker would be of little use and a combination of several biomarkers would be necessary.

ELIGIBILITY:
Inclusion Criteria:

1. age between 12 and 17 years and 11 months;
2. current clinical state of euthymia (patient stable or euthymic) after clinical evaluation, defined as the presence of clinical remission (CDRS ≤ 40, YMRS ≤ 12.5 and CGAS (Children's Global Assessment Scale) ≥ 51), being the presence of subsyndromic symptoms (YMRS> 8 and <14) admissible;
3. Presence of one or more distressing traumatic events, assessed by:

   1. Trauma subscale of the Post Traumatic Stress Disorder Questionnaire from the Schedule for Affective Disorders and Schizophrenia for School Aged Children Present and Lifetime Version (K-SADS-PL) , with frequency> 1;
   2. Holmes Rahes Stress Inventory for non-adults (H-RLSI) with frequency> 1;
   3. Children Revised Impact of Event Scale (CRIES)> 0;
   4. Childhood Trauma Questionnaire (CTQ)> 0; and
   5. at least 5 points in the disturbance assessment by the Subjective Units of Disturbance (SUDS) scale.

Exclusion Criteria:

1. substance abuse / dependence within 3 months prior to participation;
2. neurological disease or history of brain trauma;
3. autism;
4. Intelligence Quotient <70;
5. suicidal or homicidal ideation;
6. prior involvement in trauma-focused therapy;
7. psychotherapy during the study and months of follow-up, and;
8. a score greater than 25 on the Adolescent Dissociative Experience Scale, since the presence of massive dissociation requires different and more extensive treatment protocols.

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 82 (Estimated)
Dates: Start 2019-02-05 (Actual); Primary Completion 2019-08 (Estimated); Study Completion 2020-01 (Estimated)

PRIMARY OUTCOMES:
Reduction in the number of manic switches. | 12 months
  To verify if treatment with EMDR leads to a reduction in the number of manic episodes within a period of 12 months.This will be evaluated through the Young Mania Rating Scale (YMRS).
Reduction in the number of depressive episodes | 12 months
  To verify if treatment with EMDR leads to a reduction in the number of depressive episodes within a period of 12 months.This will be evaluated through the Children's Depression Rating Scale (CDRS).

SECONDARY OUTCOMES:
Change in biological markers measured by morning salivary cortisol levels in 6 months | 6 months
  To analyze the biological markers related to BD, through the measurement of morning salivary cortisol levels.
Change in biological markers measured by morning salivary cortisol levels in 12 months | 12 months
  To analyze the biological markers related to BD, through the measurement of morning salivary cortisol levels.
Change in biological markers measured by C-reactive protein levels in 6 months. | 6 months
  To analyze the biological markers related to BD, through the measurement of C-reactive protein levels.
Change in biological markers measured by C-reactive protein levels in 12 months. | 12 months
  To analyze the biological markers related to BD, through the measurement of C-reactive protein levels.
Change in biological markers measured by Brain Derived Neurotrophic Factor levels in 6 months. | 6 months
  To analyze the biological markers related to BD, through the measurement of Brain Derived Neurotrophic Factor levels.
Change in biological markers measured by Brain Derived Neurotrophic Factor levels in 12 months. | 12 months
  To analyze the biological markers related to BD, through the measurement of Brain Derived Neurotrophic Factor levels.
Change in biological markers measured by Interleukin-1 Beta levels in 6 months. | 6 months
  To analyze the biological markers related to BD, through the measurement of Interleukin-1 Beta levels.
Change in biological markers measured by Interleukin-1 Beta levels in 12 months. | 12 months
  To analyze the biological markers related to BD, through the measurement of Interleukin-1 Beta levels.
Change in biological markers measured by Interleukin-2 levels in 6 months. | 6 months
  To analyze the biological markers related to BD, through the measurement of Interleukin-2 levels.
Change in biological markers measured by Interleukin-2 levels in 12 months. | 12 months
  To analyze the biological markers related to BD, through the measurement of Interleukin-2 levels.
Change in biological markers measured by Interleukin-4 levels in 6 months. | 6 months
  To analyze the biological markers related to BD, through the measurement of Interleukin-4 levels.
Change in biological markers measured by Interleukin-4 levels in 12 months. | 12 months
  To analyze the biological markers related to BD, through the measurement of Interleukin-4 levels.
Improvement in biological markers measured by Interleukin-6 levels in 6 months. | 6 months
  To analyze the biological markers related to BD, through the measurement of Interleukin-6 levels.
Change in biological markers measured by Interleukin-6 levels in 12 months. | 12 months
  To analyze the biological markers related to BD, through the measurement of Interleukin-6 levels.
Change in biological markers measured by Interleukin-10 levels in 6 months. | 6 months
  To analyze the biological markers related to BD, through the measurement of Interleukin-10 levels.
Change in biological markers measured by Interleukin-10 levels in 12 months. | 12 months
  To analyze the biological markers related to BD, through the measurement of Interleukin-10 levels.
Change in biological markers measured by Interferon-gamma levels in 6 months. | 6 months
  To analyze the biological markers related to BD, through the measurement of Interferon-gamma levels.
Change in biological markers measured by Interferon-gamma levels in 12 months. | 12 months
  To analyze the biological markers related to BD, through the measurement of Interferon-gamma levels.
Change in biological markers measured by Tumor Necrosis Factor alpha levels in 6 months. | 6 months
  To analyze the biological markers related to BD, through the measurement of Tumor Necrosis Factor alpha levels.
Change in biological markers measured by Tumor Necrosis Factor alpha levels in 12 months. | 12 months
  To analyze the biological markers related to BD, through the measurement of Tumor Necrosis Factor alpha levels.
Modification in neurocognitive functioning through the WASI test. | 12 months
  To verify if the patients treated with EMDR will present a better profile of neurocognitive functioning, evaluated by means of the Wechsler Abbreviated Intelligence Scale (WASI).
Modification in neurocognitive functioning through the WISC-III test. | 12 months
  To verify if the patients treated with EMDR will present a better profile of neurocognitive functioning, evaluated by means of the Wechsler Intelligence Scale for Children (WISC-III) in adolescents aged up to 17 years.
Modification in neurocognitive functioning through the WAIS-III test. | 12 months
  To verify if the patients treated with EMDR will present a better profile of neurocognitive functioning, evaluated by means of the Wechsler Intelligence Scale for Adults - Third Edition (WAIS-III) for adolescents over 17 years of age.
Modification in neurocognitive functioning through the MAC Battery. | 12 months
  To verify if patients treated with EMDR will present an improvement in processing speed, access to semantic memory, and inhibitory control evaluated by means of the Verbal Fluency Tasks of the Montreal Communication Assessment Battery (MAC Battery).
Modification in neurocognitive functioning through the Hayling Test. | 12 months
  To verify if patients treated with EMDR will show an improvement in the signs of inattention, impulsivity (inhibitory failure), processing speed, semantic memory, language and cognitive flexibility through the Hayling Test.
Change in neurocognitive functioning through the MAC Battery Test. | 12 months
  To verify if patients treated with EMDR will present an improvement in short term memory, verbal work memory and inference processing through the Oral Narrative Discourse - MAC Battery test.
Change in neurocognitive functioning through the DNE test. | 12 months
  To verify if patients treated with EMDR will show an improvement in Reading Comprehension through the DNE (Discurso Narrativo Escrito or Written Narrative Speech) test.
Change in neurocognitive functioning through the NEUROPSILIN test. | 12 months
  Check if patients treated with EMDR will show an improvement in Sentence Writing (syntax) through the Spontaneous Sentence Writing Subtest - NEUPSILIN (Instrumento de Avaliação Neuropsicológica Breve Infantil or Child Brief Neuropsychological Assessment Instrument).
Change in neurocognitive functioning through the evaluation of Comprehension of Written language. | 12 months
  To verify if patients treated with EMDR will present an improvement in Comprehension of written language through the Subtest Comprehension Writing - NEUPSILIN.
Change in neurocognitive functioning through the evaluation of the Visuospatial Working Memory. | 12 months
  To verify if patients treated with EMDR will show an improvement in the Visuospatial Working Memory through the Visuospatial Working Memory Subtest - NEUPSILIN-INF.
Change in neurocognitive functioning through the Go-no-Go Subtest. | 12 months
  To verify if patients treated with EMDR will show an improvement in attention and inhibitory control through the Go-no-go Subtest - NEUPSILIN-INF.
Change in neurocognitive functioning through the Words Span in Sentences Subtest. | 12 months
  To verify if patients treated with EMDR will present an improvement in verbal work memory through the Words Span in Sentences Subtest.
Change in neurocognitive functioning through the Five Digit Test. | 12 months
  To verify if patients treated with EMDR will present an improvement in the automatic and controlled processes of attention, inhibitory control, impulsivity, self-monitoring, cognitive flexibility through the Five Digit Test.
Change in neurocognitive functioning through the Psychological Attention Battery. | 12 months
  To verify if patients treated with EMDR will show an improvement in the attention alternated, concentrated, and divided through the Psychological Attention Battery.
Change in neurocognitive functioning through the Test of School Performance. | 12 months
  To verify if patients treated with EMDR will present an improvement in the school performance in writing of words in reading, writing of isolated words and arithmetic through the Test of School Performance.

CONTACTS AND LOCATIONS:
Overall Officials: Ives C Passos, PhD, Principal Investigator — Federal University of Health Science of Porto Alegre
Locations (1):
- Centro de Pesquisas Clínicas do Hospital de Clínicas de Porto Alegre, Porto Alegre, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: Undecided